CLINICAL TRIAL: NCT04875286
Title: Patient Reported Symptom Control With THC or CBD Use
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-0753; NCI-2021-02853 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0753 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-04-22; First posted 2021-05-06 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Cancer-Associated Pain; Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Cancer Pain; Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (medical record review, questionnaires)): Patients' medical records are reviewed and then complete questionnaires over 27 minutes.
  Interventions: Other: Electronic Health Record Review; Other: Questionnaire Administration

INTERVENTIONS:
Other: Electronic Health Record Review — Medical records reviewed
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study compares patients' attitudes regarding marijuana products for medical use and other treatments for cancer-related pain. This study may help researchers gain better understanding of patient's perception on their use of marijuana products in treating cancer-related pain and other common cancer-related symptoms.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the patient's reported preference for cancer pain improvement with opioids, opioids with delta-9-tetrahydrocannabinol (THC)-marijuana and/or opioids with cannabidiol (CBD).

SECONDARY OBJECTIVES:

I. To determine the association between perception of cancer-related symptom relief and use of THC-marijuana and/or CBD.

II. To compare patient perception of THC-marijuana and/or CBD versus (vs.) cancer treatments in treatment of cancer.

III. To evaluate patient report of adverse effects experienced while using THC-marijuana and/or CBD.

IV. To evaluate patient reported concerns while using THC-marijuana and/or CBD. V. To evaluate patient attitude of dosing, forms and use of THC-marijuana and/or CBD.

VI. To evaluate demographic, physical and psychosocial factors that influence patient perception and attitudes of THC-marijuana and/or CBD.

VII. To explore the difference of patient perception of THC-marijuana and CBD in cancer centers in a legalized vs. a non-legalized state.

VIII. To explore the patient reported preference of THC-marijuana and CBD for cancer pain and symptom relief of patients in a Supportive Care Center vs. Integrative Medicine Center at University of Texas (U.T.) MD Anderson.

OUTLINE:

Patients' medical records are reviewed and then complete questionnaires over 27 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Patients (inpatient or outpatient) seen by the Palliative Care and Integrative Medicine teams at The University of Texas MD Anderson Cancer Center (Texas) and the Palliative Care team at Banner MD Anderson Cancer Center (Arizona)
* Patients must be primary residents of Texas or Arizona
* Patients able to speak and read English
* Patients are 18 years old and above
* Patients should have a cancer diagnosis, cancer-associated pain, and taking strong opioids (morphine, oxycodone, hydrocodone, hydromorphone, oxymorphone, methadone, fentanyl)
* Patients who have used in the past 3 months or are using alternative botanical pain management while under prescription opioids

Exclusion Criteria:

* Patients who are not able to speak or read English
* Altered mental status as determined by the interviewer based on the ability to understand the nature of the study and consent process
* Patients who have not used medical marijuana and/or CBD products
* Patients who do not have cancer
* Patients who do not have cancer-associated pain
* Patients who are not taking opioids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients (inpatient or outpatient) seen by the Palliative Care and Integrative Medicine teams at The University of Texas MD Anderson Cancer Center (Texas) and the Palliative Care team at Banner MD Anderson Cancer Center (Arizona)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who prefer opioids with THC-marijuana and/or opioids with cannabidiol (CBD) to opioids alone for their cancer pain relief | through study completion, an average of 1 year
  Will be calculated and reported along with a 95% confidence interval.

SECONDARY OUTCOMES:
Perception of cancer-related symptom relief | through study completion, an average of 1 year
  Will be associated with use of THC-Marijuana and/or CBD. Will be evaluated by generalized linear mixed models to account for the dependency among those patients who have used/are using both.
Patient perception of THC-marijuana and/or CBD | through study completion, an average of 1 year
  Compared to cancer treatments in treatment of cancer. Will be evaluated by generalized linear mixed models to account for the dependency among those patients who have used/are using both.
To evaluate patient report of adverse effects experienced while using THC-marijuana and/or CBD | through study completion, an average of 1 year
  Patient reported outcomes will be summarized by frequency and proportion.
To evaluate patient reported concerns while using THC-marijuana and/or CBD | through study completion, an average of 1 year
  Patient reported outcomes will be summarized by frequency and proportion.
Patient attitude of dosing, forms and use of THC-marijuana and/or CBD | through study completion, an average of 1 year
  Patient reported outcomes will be summarized by frequency and proportion.
Demographic, physical and psychosocial factors that influence patient perception and attitudes of THC-marijuana and/or CBD | through study completion, an average of 1 year
  Will be evaluated by Wilcoxon rank sum (Kruskal-Wallis) test or chi-square (Fisher's exact) test, when appropriate. To further evaluate these associations, univariate and multivariable logistic regression models will be fitted. Multiple comparisons will be adjusted where appropriate.
To explore the difference of patient perception of THC-marijuana and CBD in cancer centers in a legalized vs. a non-legalized state. | through study completion, an average of 1 year
  Differences will be explored.
Patient reported preference of THC-Marijuana and CBD for cancer pain and symptom relief of patients | through study completion, an average of 1 year
  Will be explored between a Supportive Care Center vs. Integrative Medicine Center at University of Texas (U.T.) MD Anderson. Will be evaluated by Wilcoxon rank sum (Kruskal-Wallis) test or chi-square (Fisher's exact) test, when appropriate. To further evaluate these associations, univariate and multivariable logistic regression models will be fitted. Multiple comparisons will be adjusted where appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberson C Tanco, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - M D Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org